CLINICAL TRIAL: NCT02113501
Title: Optimized Treatment Strategy for HighGradeT1 (HGT1) Bladder Cancer Based on Substaging (Depth of Lamina Propria Invasion): a Prospective Observational Cohort Study
Brief Title: Optimized Treatment Strategy for HighGrade1 (HGT1) Bladder Cancer Based on Substaging: a Prospective Observational Cohort Study
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HighGradeT1 Bladder Cancer HVH
Record Dates: First submitted 2014-03-31; First posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Bladder Cancer
Keywords: HGT1; high risk bladder cancer; substaging; repeat transurethral resection (reTUR); lamina propria
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — paraffin embedded blocks of transurethral resection (TUR) samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HGT1a: HGT1a bladder cancer patients will undergo BCG induction and maintenance followed by conventional follow-up (cystoscopy and cytology at 3months and then every 6months).
- HGT1b: HGT1b bladder cancer patients will undergo a 2nd TUR after BCG induction. If negative, continue with maintenance BCG followed by conventional follow-up (cystoscopy and cytology every 6months).

SUMMARY:
Non-muscle invasive bladder cancer of High Grade stage T1 (HGT1), has up to 20% risk of progression to invasive disease. Because the depth of substaging seems to identify two separate groups with different progression risk (HighGradeT1a and HighGradeT1b), we design a differential treatment strategy for each group. The main hypothesis is that HighGradeT1a bladder cancer can spare a second endoscopic procedure.

DETAILED DESCRIPTION:
Only cases of initial diagnosis of HighGradeT1 and with a complete transurethral endoscopic resection (TUR) of bladder tumor) can enter this protocol. HighGradeT1a will only receive standard BCG treatment (induction and maintenance). HighGradeT1b will undergo a second transurethral endoscopic resection (TUR) after the induction of Bacillus de Calmette-Guerin (BCG) and then continue mantenaince BCG and standard follow-up.

ELIGIBILITY:
Inclusion Criteria:

* HGT1 bladder cancer at initial diagnosis and after a complete TUR

Exclusion Criteria:

* abscence of muscularis propria in the TUR specimen

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Initial HGT1 bladder cancer patients that have undergone a complete TUR and are willing to enter the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2005-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
progression | 5year

SECONDARY OUTCOMES:
recurrence | 5year

OTHER OUTCOMES:
Cancer specific survival | 5year

CONTACTS AND LOCATIONS:
Overall Officials: Anna Orsola, MD, Principal Investigator — Hospital Vall d'Hebron, Barcelona, Spain
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain, Barcelona, Barcelona, Spain

REFERENCES:
- [Result] Orsola A, Cecchini L, Raventos CX, Trilla E, Planas J, Landolfi S, de Torres I, Morote J. Risk factors for positive findings in patients with high-grade T1 bladder cancer treated with transurethral resection of bladder tumour (TUR) and bacille Calmette-Guerin therapy and the decision for a repeat TUR. BJU Int. 2010 Jan;105(2):202-7. doi: 10.1111/j.1464-410X.2009.08694.x. Epub 2009 Jun 24. PMID 19558557